CLINICAL TRIAL: NCT00150787
Title: A Multicenter, Double-blind, Follow-up Trial Evaluating the Long-term Safety of Levetiracetam (1000 to 3000 mg/Day Oral b.i.d.) and Carbamazepine (400 to 1200 mg/Day Oral b.i.d.), Used as Monotherapy in Subjects (≥ 16 Years) Coming From the N01061 Trial.
Brief Title: Monotherapy With Levetiracetam or Carbamazepine in Patients Suffering From Epilepsy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01093
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy, Tonic-clonic
Keywords: Monotherapy, epilepsy; Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: LEVETIRACETAM

SUMMARY:
A double-blind follow-up trial assessing the long term safety of Levetiracetam as per adverse events reporting, physical and neurological examination and vital signs

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis of epilepsy.
* Subjects having experienced in the past unprovoked partial seizures (IA, IB, IC with clear focal origin), or generalized tonic-clonic seizures (without clear focal origin), that are classifiable according to the International Classification of Epileptic Seizures
* Subjects coming from the N01061 monotherapy trial and for whom double-blind continuation of investigational product is beneficial.

Exclusion Criteria:

* Need for an additional AED.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2003-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Around 2 years of Safety assessment of levetiracetam via Adverse Events reporting, physical and neurological examination and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Brodie MJ, Perucca E, Ryvlin P, Ben-Menachem E, Meencke HJ; Levetiracetam Monotherapy Study Group. Comparison of levetiracetam and controlled-release carbamazepine in newly diagnosed epilepsy. Neurology. 2007 Feb 6;68(6):402-8. doi: 10.1212/01.wnl.0000252941.50833.4a. PMID 17283312